CLINICAL TRIAL: NCT01885234
Title: Aerobic Training Effect in Pregnant Women With Gestational Diabetes and Chronic Hypertension: Randomized Clinical Trial
Brief Title: Aerobic Training in Pregnant Women With Gestational Diabetes and Chronic Hypertension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: GDM-HAS120008
Record Dates: First submitted 2013-06-05; First posted 2013-06-24 (Estimated); Last update posted 2015-12-22 (Estimated); Status verified 2015-12

CONDITIONS: Pregnancy; Gestational Diabetes Mellitus; Chronic Hypertension in Obstetric Context
Keywords: Glycated hemoglobin; HOMA; Pregnancy; aerobic exercise
MeSH Terms: conditions — Diabetes, Gestational | interventions — Exercise; Plyometric Exercise

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Aerobic exercise (Experimental): Pregnant women with Gestational Diabetes and pregnant women with chronic hypertension will perform 50 minutes of aerobic exercise in a bicycle, 3 times a week
  Interventions: Other: Aerobic exercise
- Stretch exercise (Placebo Comparator): Pregnant women with Gestational Diabetes and pregnant women with chronic hypertension will perform 50 minutes of stretch exercise, once a week
  Interventions: Other: Stretch exercise

INTERVENTIONS:
Other: Aerobic exercise — Pregnant women with Gestational Diabetes and pregnant women with chronic hypertension will perform 50 minutes of aerobic exercise in a bicycle, 3 times a week
  Arms: Aerobic exercise
Other: Stretch exercise — Pregnant women with Gestational Diabetes and pregnant women with chronic hypertension will perform 50 minutes of stretch exercise, once a week
  Arms: Stretch exercise

SUMMARY:
The aim of the present study is verify glycated hemoglobin (HbA1c) and HOMA behavior in pregnant women with gestational diabetes or chronic hypertension after an aerobic training in cycle-ergometer. The sample is composed by 64 pregnant and sedentary women, 20 weeks' pregnant.

Two experimental groups (gestational diabetes and chronic hypertension, n = 16 each) will perform a low-intensity aerobic training in cycle-ergometer, three times/week, for 45 minutes each session. Two control groups (gestational diabetes and chronic hypertension, n = 16 each) will perform an unique session/week of relaxation and stretching.

Outcomes: first ventilatory threshold, HbA1c,HOMA, type of delivery, weight and height of the newborn.

DETAILED DESCRIPTION:
The statistical analysis will consist of:

* descriptive statistic;
* Levene's test
* Shapiro Wilk's normality test
* Parametric or non-parametric test
* a=0.05
* SPSS 17.0

ELIGIBILITY:
Inclusion Criteria:

* age > 20 years;
* gestational age between 20 and 27 weeks (date of the last period and confirmed by ultrasound);
* Only one foetus in the womb;
* Without orthopedic limitations;
* Non-smoker;
* Medical clearance for exercise

Exclusion Criteria:

* Pre-eclampsia;
* fetal malformations;
* Intrauterine fetal death

Ages: 20 Weeks to 27 Weeks | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 9 (Actual)
Dates: Start 2011-12; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
glycated hemoglobin | day 1 and 10 weeks after training

SECONDARY OUTCOMES:
HOMA | day 1 and 10 weeks after training

OTHER OUTCOMES:
First ventilatory threshold | day 1 and 10 weeks after training

CONTACTS AND LOCATIONS:
Overall Officials: José Geraldo L Ramos, MD, Principal Investigator — HC Porto Alegre
Locations (1):
- Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil